CLINICAL TRIAL: NCT02277093
Title: Phase II Study With Pacritinib to Inhibit JAK/STAT Signaling in Refractory Colorectal Cancer
Brief Title: Pacritinib to Inhibit JAK/STAT Signaling in Refractory Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA issued a clinical hold as pacritinib had increased side effects
Sponsor: Washington University School of Medicine (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201412087
Record Dates: First submitted 2014-10-24; First posted 2014-10-28 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pacritinib (Experimental): * Pacritinib is an oral drug which will be taken on an outpatient basis daily on a 28-day cycle at a dose of 200 mg twice a day (BID)
  * Pacritinib should be take at approximately the same times every day with a glass of water, with or without food
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib
  Other Names: SB1518

SUMMARY:
The investigators propose to assess the efficacy, progression-free survival, and adverse events of pacritinib in patients with refractory colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed refractory colorectal cancer
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with CT scan, as >20 mm by chest x-ray, or >10 mm with calipers by clinical exam.
* Refractory to or intolerant of standard systemic therapy, including having received two or more standard available therapies known to prolong survival for which s/he was eligible, including FOLFOX or FOLFIRI with or without bevacizumab, aflibercept, cetuximab, or panitumumab
* At least 18 years of age.
* ECOG performance status < 2
* Life expectancy ≥ 12 weeks.
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 50,000/mcl
  * Total bilirubin ≤ 2.0 x IULN
  * AST (SGOT) / ALT (SGPT) ≤ 3.0 x IULN
  * Serum creatinine ≤ 2.0 mg/dL OR creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above 2.0 mg/dL
  * Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
  * Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior therapy with a JAK2 or FLT3 inhibitor.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Received any chemotherapeutic or targeted agent for metastatic colorectal cancer within two weeks of initiation of study drug.
* Currently receiving any other investigational agents.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pacritinib or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with pacritinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Use of potent cytochrome P450 3A4 (CYP3A4) inhibitor within one week of pacritinib initiation.
* Patients with CTCAE grade 2 cardiac arrhythmias may be considered for inclusion if the arrhythmias are stable, asymptomatic, and unlikely to affect patient safety. Patients will be excluded if they have ongoing cardiac dysrhythmias of CTCAE grade ≥ 3, corrected QT interval (QTc) prolongation >450ms, or other factors that increase the risk for QT interval prolongation (eg, heart failure, hypokalemia [defined as serum potassium <3.0mEq/L that is persistent and refractory to correction], or family history of long QT interval syndrome).
* Any gastrointestinal (GI) or metabolic condition that could interfere with absorption of oral medication such as ongoing grade 3 or higher diarrhea, constipation, nausea, or vomiting.
* Active viral hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin R Tan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pacritinib
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pacritinib
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 63 [43 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 11
Primary Site of Cancer [Count of Participants; unit: Participants]
  Right colon | 7
  Left colon | 2
  Rectal | 2
Baseline c-reactive protein (CRP) [Median (Full Range); unit: mg/L] — Population: 2 out of the 11 patients did not have a baseline c-reactive protein.
  mg/L
    number analyzed (Participants) | 9
    (all) | 12.1 [2.1 to 147]
Prior lines of therapy for metastatic disease [Median (Full Range); unit: prior lines of therapy] | 4 [2 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  Progression - at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Through completion of follow-up (median follow-up was 6.61 months)
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Pacritinib
Number analyzed (Participants) | 11
months | 1.91 [1.81 to 8.75]

2. Secondary Outcome: Toxicity Profile and Tolerability as Measured by Reportable Adverse Events
Description: * The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
  * Reportable adverse events will be tracked for 28 days following the last day of study treatment. For the purposes of this protocol, reportable adverse events are events that are greater than or equal to grade 2 and are considered possibly, probably, or definitely related to study treatment.
Time Frame: Up to 28 days following last day of study treatment
Measure: Number; unit: adverse event
Arm/Group | Pacritinib
Number analyzed (Participants) | 11
adverse event
  Diarrhea | 1
  Edema limbs | 1
  Edema face | 1
  Fatigue | 1
  Localized edema | 1
  Blood bilirubin increased | 1
  Dyspnea | 1
  Rash maculopapular | 1

3. Secondary Outcome: Overall Response Rate (ORR)
Description: * The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
  * Using RECIST 1.1
  * The follow-up time was calculated from the start of treatment until death or on the final collection date of data on 10/27/2016.
Time Frame: Through completion of follow-up (median follow-up was 6.61 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib
Number analyzed (Participants) | 11
Participants
  Complete response | 0
  Partial response | 0
  Stable disease | 1
  Progressive disease | 6
  Not evaluable | 4

4. Secondary Outcome: Time to Progression (TTP)
Time Frame: Through completion of follow-up (median follow-up was 6.61 months)
Population: Only patients who had their first measurement scans were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Pacritinib
Number analyzed (Participants) | 7
months | 1.73 (0.26)

5. Secondary Outcome: Overall Survival (OS)
Description: -The follow-up time for OS was calculated from the start of treatment until death or on the final collection date of data on 10/27/2016.
Time Frame: Through completion of follow-up (median follow-up was 6.61 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pacritinib
Number analyzed (Participants) | 11
months | 6.61 [2.79 to 9.34]

ADVERSE EVENTS:
Arm/Group | Pacritinib
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pacritinib (N=11)
Alkaline phosphatase increased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Platelet count decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pacritinib (N=11)
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Rectal pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Abdominal cramps (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Edema limbs (General disorders) | 2
Edema face (General disorders) | 1
Fatigue (General disorders) | 3
Localized edema (General disorders) | 1
Anorectal infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Please note that the study ended early due to the FDA issuing a clinical hold as pacritinib had increased side effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes